CLINICAL TRIAL: NCT04565834
Title: Étude Des Altérations Génétiques (polymorphismes) Des Gènes-clés De La Voie Kynurénine Sur Le Comportement Suicidaire
Brief Title: Effect of Genetic Alterations Affecting the Genes Encoding the Major Enzymes of the Kynurenine Pathway on Suicidal Behavior
Acronym: SuiKYN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Universidad Autonoma de Madrid (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2019-2/JLC-01
Record Dates: First submitted 2020-09-14; First posted 2020-09-25 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2023-06

CONDITIONS: Tryptophan Metabolism Alterations; Polymorphism; Suicidal Behavior
Keywords: sucidal behavior; Inflammation; Kynurenines
MeSH Terms: conditions — Inflammation | interventions — Polymorphism, Single Nucleotide; Genotype

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — These are biological samples collected from previous registered studies (SUI-PREDICT, SMART CRISIS, SPAD) as well as samples from the Human Molecular Genetics Laboratory A-209 from the Faculty of Biology at the Independent University of Madrid, Spain.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- : Suicide attempters: 325 patients who have made at least one attempt to commit suicide.
  Interventions: Genetic: SNP (single nucleotide polymorphism) genotyping
- Depressed non-attempters: 99 patients suffering from depression but have never attempted to commit suicide.
  Interventions: Genetic: SNP (single nucleotide polymorphism) genotyping
- Healthy controls: 425 healthy subjects (i.e. those who have no mental disorders and have never attempted to commit suicide)
  Interventions: Genetic: SNP (single nucleotide polymorphism) genotyping

INTERVENTIONS:
Genetic: SNP (single nucleotide polymorphism) genotyping — We use TaqMan technique to perform SNP genotyping. The PCR reactions are carried out using the Roche "Light Cycler 480" thermal cycler following the protocol recommended by Thermo Fisher Scientific. Then, replication of 10% of the samples is carried out.
  Other Names: Determination of allelic and genotypic frequencies of IDO1 rs7820268, IDO2 rs10109853, KMO rs1053230, KAT1 rs10988134 and ACMSD rs2121337 SNPs in each group

SUMMARY:
Current research has shown that an imbalance in the Kynurenine pathway plays a role in the physiopathology of neurogenerative and mental disorders (with a decrease in neuroprotective metabolites and an increase in neurotoxic products). So far the research has concentrated on the enzymes IDO 1/2, KAT (1-4), KMO and ACMSD which are the key players in this pathway. Several polymorphisms affecting these enzymes have been associated with certain disorders characterized by a deregulation of the inflammation and immune response (McCauley et al 2009,Tardito et al 2013, Lee et al 2014), but the link between these enzymes and suicidal behavior is not yet clear. The investigators hypothesize that people with history of suicide attempt would have a genetic alterations of the kynurenine pathway specific for suicidal behavior.

ELIGIBILITY:
Inclusion Criteria:

* For the "Sucide attempters" group: Any patient aged 18 or over who has made at least one suicide attempt.
* For the two control groups: Any patient aged 18 or over, suffering from depression but has never attempted to commit suicide and any healthy subject who has never had any mental disorders.

Exclusion Criteria:

* Any patient who has expressed opposition to the use of his/her data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients for whom biological samples have been collected and registered in the hospital's databank for the purpose of previously registered studies : SPAD (RCB no. 2016-A01375-46), SMART-CRISIS (RCB no.: 2017-A02634-49) and SUI-PREDICT (RCB no.: 2016-A00845-46) and several studies conducted at the university hospitals of Puerta de Hierro, Ramon y Cajal et Fundacion Jiminez Diaz in Madrid, Spain, since 2004.
Sampling Method: Non-Probability Sample
Enrollment: 849 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
The genotypic and allelelic frequencies of IDO1 rs7820268 SNP in each studied group | 24 months
  The frequencies of this SNP will be measured as a percentage
The genotypic and allelelic frequencies of IDO2 rs10109853 SNP in each studied group | 24 months
  The frequencies of this SNP will be measured as a percentage
The genotypic and allelelic frequencies of KMO rs1053230 SNP in each studied group | 24 months
  The frequencies of this SNP will be measured as a percentage
The genotypic and allelelic frequencies of KAT1 rs10988134 SNP in each studied group | 24 months
  The frequencies of this SNP will be measured as a percentage
The genotypic and allelelic frequencies of ACMSD rs2121337 SNP in each studied group | 24 months
  The frequencies of this SNP will be measured as a percentage

OTHER OUTCOMES:
Age of subjects | 24 months
  The age will be recorded for statistical purposes
Gender of subjects | 24 months
  The gender will be recorded for statistical purposes
Marital status of subjects | 24 months
  The marital status will be recorded as a number and a percentage
Education level of subjects | 24 months
  the education level will be recorded as a number and a percentage
Diagnosis | 24 months
  The diagnosis will be recorded as a number and a percentage
Number of suicide attempts | 24 months
  The number of suicide attempts will be recorded as a number
Age of first suicide attempt | 24 months
  Age of first suicide attempt will be recorded as a number

CONTACTS AND LOCATIONS:
Locations (2):
- Department of Psychiatry, Nimes University Hospital, Nîmes, Gard, France
- José-Fernandez-Piqueras, Madrid, Spain